CLINICAL TRIAL: NCT06847308
Title: Visual Biofeedback (VB) Through Trans-Perineal Ultrasound (TPU) During the Active 2nd Stage of Labour to Improve Maternal Childbirth Satisfaction: a Randomised Controlled Trial
Brief Title: Visual Biofeedback Through Transperineal Ultrasound During the Expulsive Phase of Labour to Improve Maternal Childbirth Satisfaction
Acronym: RCT:VB-TPU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S68276; 1S49923N (Other Grant/Funding Number: Research Council Flanders (FWO))
Record Dates: First submitted 2024-12-05; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Labor Stage, Second; Labor and Delivery; Satisfaction With Care; Childbirth
Keywords: 2nd stage of labour; visual biofeedback; maternal childbirth satisfaction; obstetrics; ultrasound; trans-perineal ultrasound
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Trial statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - VB with TPUS (Active Comparator): Use of ultrasound for visual biofeedback
  Interventions: Behavioral: visual biofeedback through trans-perineal ultrasound
- Control Group - standard of care (No Intervention): Control group that will receive standard of care

INTERVENTIONS:
Behavioral: visual biofeedback through trans-perineal ultrasound — Trans-perineal ultrasound will be used to provide visual biofeedback during the active 2nd stage of labour, this for ten consecutive uterine contractions / pushing efforts
  Arms: Intervention - VB with TPUS

SUMMARY:
Childbirth is generally regarded as a positive life-changing experience. Up to 44% of women may however experience this as a traumatic event, with 3% suffering from post-traumatic stress disorder after childbirth. The aetiology of a traumatic childbirth experience is a complex interplay between pre-birth, intra-partum and postnatal factors. Feelings of loss of control, lack of interaction with the obstetric caregiver and lack of emotional or practical support during labour are important contributing factors. This trial aims to investigate the effect of providing Visual Biofeedback (VB) through Trans-Perineal Ultrasound (TPU) during the active 2nd stage of labour on maternal childbirth satisfaction. The hypothesis is that the intervention will improve patient-caregiver communication and enhance parturient women's sense of control and empowerment, ultimately improving the birth experience.

ELIGIBILITY:
INCLUSION criteria (all must be met):

1. Voluntary written informed consent of the participant.
2. Term (37-42w) singleton gestations.
3. Vaginally nulliparous (no previous vaginal birth > 20 weeks of gestation).
4. Fetus in cephalic presentation, without any major congenital or chromosomal anomalies.
5. Admitted to the delivery unit in labour, regardless of the onset (spontaneous or induced).
6. Epidural analgesia in situ.
7. Non-pathological CTG at the time of recruitment (2015 FIGO classification).

EXCLUSION criteria (if one or more is present):

* Significant psychiatric comorbidity (psychiatric follow-up during pregnancy, or active (psycho-pharmacological) treatment).
* History of severe PFDs/surgery (or any other condition affecting pelvic floor function/anatomy, besides pregnancy and delivery).
* Significant neurological disease e.g., spinal injury, multiple sclerosis, diabetic neuropathy, etc.
* Significant connective tissue disorders (e.g., Ehlers-Danlos syndrome).
* Severe active maternal (pregnancy-related) comorbidity: non-exhaustive e.g., severe hypertensive disorder, significant antepartum haemorrhage, sepsis, thromboembolism, severe pre-existing cardiac/respiratory/neurological disease, etc. Well-controlled comorbidities will not be considered exclusion criteria (non-exhaustive e.g., well-controlled (gestational) diabetes, hypertensive disorders of pregnancy, PROM without signs of intra-amniotic infection, etc.).
* Linguistic barriers - not able to give written informed consent in Dutch.
* Severe visual impairment (sufficient to the receipt/comprehension of visual biofeedback).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-03 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Maternal childbirth satisfaction | From enrollment to two days after delivery
  Maternal childbirth satisfaction will be assessed using the Birth Satisfaction Scale revised (BSS-R) questionnaire. The total score ranges from 0/40 to 40/40, with lower scores indicating worser satisfaction.
Vaginal birth-induced perineal trauma | Assessment immediately after childbirth (delivery of the baby)
  Assessed immediately after delivery through clinical examination (inspection and palpation) of the perineal region and grading of any injury according to the Sultan classification (intact - firs degree tear: vaginal mucosa/perineal skin - second degree tear: perineal muscles - third degree tear: external and/or internal anal sphincter - fourth degree tear: anorectal mucosa).

SECONDARY OUTCOMES:
Delivery mode | From enrollment to the end of the delivery
  Spontaneous vaginal vs. operative delivery (vacuum and/or forceps delivery or 2nd stage caesarean section).
Urinary incontinence | From enrollment to the end of follow-up at 1 year postpartum
  The presence and severity of urinary incontinence will be assessed twice: once around 12 weeks postpartum, and once additionally 6-12 months postpartum. The incidence and severity of urinary incontinence will be self-reported, using the standardized and validated International Consultation on Incontinence Questionnaire - Short Form questionnaire for urinary incontinence. Total scores range from 0/21-21/21, with higher scores indicating worser symptoms.
Anal incontinence | From enrollment to the end of follow-up at 1 year postpartum
  The presence and severity of anal incontinence will be assessed twice: once around 12 weeks postpartum, and once additionally 6-12 months postpartum. The incidence and severity of anal incontinence will be self-reported, using the standardized and validated St. Marks Incontinence Score. Total scores range from 0/24-24/24, with higher scores indicating worser symptoms.
Prolapse symptoms | From enrollment to the end of follow-up at 1 year postpartum
  The presence and severity of prolapse symptoms will be assessed twice: once around 12 weeks postpartum, and once additionally 6-12 months postpartum. The incidence and severity of prolapse symptoms will be self-reported, using the standardized and validated Pelvic Organ Prolapse Distress Index for symptoms of pelvic organ prolapse. Total scores range from 0/24-24/24, with higher scores indicating worser symptoms.
Sexual function | From enrollment to the end of follow-up at 1 year postpartum
  Sexual function will be assessed twice: once around 12 weeks postpartum, and once additionally 6-12 months postpartum. Sexual function will be self-reported, using the standardized and validated Female Sexual Function Index (19 items, range 2/36-36/36). Higher scores indicate more severe dysfunction.
Sexual function | From enrollment to the end of follow-up at 1 year postpartum
  Sexual function will be assessed twice: once around 12 weeks postpartum, and once additionally 6-12 months postpartum. Sexual function will be self-reported, using the standardized and validated Female Sexual Distress Scale-Revised questionnaire (13 items, range 0/52-52/52). Higher scores indicate more severe dysfunction.
Duration of the total second stage | From the onset of full cervical dilatation (= onset of the second stage) until childbirth (= delivery of the baby), estimated to range between 0-180 minutes.
  The period between full cervical dilatation and delivery of the baby.
Duration of the active total second stage | From the onset of active maternal pushing efforts (= onset of the active second stage) and childbirth (= delivery of the baby), estimated to range between 0-120 minutes.
  The period between the onset of active maternal pushing efforts (= active second stage) and delivery of the baby.
Delta-AoP | During the active second stage of labour, from the first to the 10th consecutive pushing effort, estimated interval 20 minutes (4-5 contractions/10 minutes).
  Differences in the angle of progression (AoP, in degrees) at rest and maximal Valsalva during the active 2nd stage (i.e., active maternal pushing efforts), measured by transperineal ultrasound during the first and 10th consecutive pushing effort.
Delta LAM | During the active second stage of labour, from the first to the 10th consecutive pushing effort, estimated interval 20 minutes (4-5 contractions/10 minutes).
  Differences in the anteroposterior diameter of the puborectalis part of the levator ani muscle (LAM) at rest and maximal Valsalva during the active 2nd stage (= active maternal pushing efforts), measured by transperineal ultrasound during the first and 10th consecutive pushing effort.

CONTACTS AND LOCATIONS:
Overall Officials: Jute Richter, MD, PhD, Principal Investigator — University Hospitals Leuven / KU Leuven; Jan Deprest, MD, PhD, Principal Investigator — University Hospitals Leuven / KU Leuven
Locations (1):
- The University Hospitals Leuven, Leuven, Vlaams-Braband, Belgium

IPD SHARING:
Plan to Share IPD: No
Privacy and ethical restrictions